CLINICAL TRIAL: NCT06557733
Title: Phase 2 Study to Evaluate the Efficacy and Safety of TPST-1495 in Patients With Familial Adenomatous Polyposis (FAP)
Brief Title: An Investigational Drug (TPST-1495) in Patients With Familial Adenomatous Polyposis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2024-06758; NCI-2024-06758 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UWI23-16-01 (Other: University of Wisconsin Carbone Cancer Center - University Hospital); UWI23-16-01 (Other: DCP); P30CA014520 (NIH); UG1CA242596 (NIH); UG1CA242635 (NIH)
Record Dates: First submitted 2024-08-15; First posted 2024-08-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Familial Adenomatous Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Biopsy; Specimen Handling; Endoscopy, Digestive System; Gastroscopy; Endoscopy, Gastrointestinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (TPST-1495) (Experimental): Patients receive TPST-1495 PO QD for 6 months in the absence of unacceptable toxicity. Patients also undergo EGD and GI endoscopy with biopsy at baseline and end of treatment and undergo blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: EP2/EP4 Antagonist TPST-1495; Procedure: Esophagogastroduodenoscopy; Procedure: Gastrointestinal Endoscopy; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: EP2/EP4 Antagonist TPST-1495 — Given PO
  Other Names: Dual EP2/4 Antagonist TPST-1495; PGE2 EP2/EP4 Receptor Antagonist TPST-1495; Prostaglandin E2 Receptor EP2/EP4 Antagonist TPST-1495; TPST 1495; TPST-1495; TPST1495
Procedure: Esophagogastroduodenoscopy — Undergo EGD
  Other Names: EGD; Upper Endoscopy
Procedure: Gastrointestinal Endoscopy — Undergo GI endoscopy
  Other Names: Enteroscopy
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This open-label phase II trial tests how well TPST-1495 works in reducing the number of polyps in the small bowel and colon in patients with familial adenomatous polyposis (FAP). FAP is an inherited condition in which numerous polyps (growths that protrude from mucous membranes) form on the inside walls of the colon and rectum. It increases the risk for colon cancer. TPST-1495 binds to specific prostaglandin receptors. TPST-1495 is a dual antagonist of the prostaglandin E2 (PGE2) receptor subtypes EP2 and EP4, while sparing the immune-stimulating EP1 and EP3 receptors. TPST-1495 may help reduce the number of polyps in the small bowel and colon in patients with FAP.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of TPST-1495 in reducing duodenal polyp burden in patients with FAP.

II. To assess the safety of TPST-1495 in patients with FAP; we will evaluate the incidence of grade 2 or 3 adverse events.

SECONDARY OBJECTIVE:

I. The activity of TPST-1495 in reducing rectum/IPAA (ileal pouch-anal anastomosis) polyp burden in patients with FAP.

EXPLORATORY OBJECTIVES:

I. Reduction in intestinal polyp burden as a function of immunohistochemical staining at baseline and end of intervention (6-months) of rectal and duodenal tissue samples for COX-2 expression level, beta-catenin, and Ki-67.

II. Proteomic profile of serum correlated to clinical response to therapy compared between baseline and end of intervention.

III. Biospecimen acquisition. IV. TPST-1495 concentrations in plasma at pre-dose, 2-, and 4-hours post-dose at month 3 visit to assess steady-state pharmacokinetics.

OUTLINE:

Patients receive TPST-1495 orally (PO) once daily (QD) for 6 months in the absence of unacceptable toxicity. Patients also undergo esophagogastroduodenoscopy (EGD) and gastrointestinal (GI) endoscopy with biopsy at baseline and end of treatment and undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of familial adenomatous polyposis (FAP), defined as at least one of the following:

  * Genetic diagnosis with confirmed APC mutation (clinical CLIA [clinical laboratory improvement amendments] certified lab or research testing)
  * Obligate carrier
  * Clinical diagnosis of classic FAP with ≥ 100 colorectal adenomas status post colectomy and a family history of FAP
  * Clinical diagnosis of FAP, based on personal and family history. Note: This criterion requires documented review and agreement from either the study chair or the MW consortium lead investigator
* Previously underwent prophylactic colectomy with IRA (ileo-rectal anastomosis) or IPAA at least 12 months before pre-registration evaluation and without ongoing surgical complication
* Willing to discontinue taking non-steroidal anti-inflammatory drugs (NSAIDs) 5 days prior to initiation of study treatment and limit frequency of NSAID dosing during study treatment
* Age ≥ 18. Because no dosing or adverse event (AE) data are currently available on the use of TPST-1495 in participants < 18 years of age, children and adolescents are excluded from this study but will be eligible for future pediatric trials, if applicable
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Leukocytes (white blood count [WBC]) ≥ 3,000/uL (≥ 2,500/uL for African American participants)
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 11.5 g/dL
* Total bilirubin ≤ 1.5 x institutional upper limit normal (ULN) (unless patient has Gilbert's)
* Alkaline phosphatase ≤ 1.5 x institutional ULN
* Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) ≤ 2 x institutional ULN
* Alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) ≤ 2 x institutional ULN
* Creatinine ≤ institutional ULN
* Urinary testing results within institutional limits of normal or deemed clinically insignificant
* Patients on chronic suppressive antiviral therapy for herpes simplex virus (HSV) are eligible
* Presence of Spigelman 2 or 3 duodenal polyposis stage assessed by endoscopy
* Not pregnant: The effects of TPST-1495 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation including 90 days after discontinuing study agent. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Not currently breastfeeding
* Ability to understand and the willingness to sign a written informed consent document
* Helicobacter (H.) pylori negative confirmed with gastric biopsy (at time of screening EGD). If positive for H. pylori the patient can be offered full course of approved therapy with confirmation of eradication and re-assessment for trial participation with likely need to repeat baseline endoscopies if > 45 days since date of baseline procedures

Exclusion Criteria:

* Use of any other investigational agents ≤ 12 weeks prior to pre-registration
* History of gastric or intestinal ulceration due to NSAID therapy
* Uncontrolled intercurrent illness or recent surgical procedure that in the opinion of the investigative team would limit compliance with study requirements
* History of invasive malignancy ≤ 3 years prior to pre-registration (exception: adequately treated carcinoma of the cervix, carcinoma in situ, or basal or squamous cell carcinomas of the skin)
* History of any upper GI surgery that does not permit access to or evaluation of a 10 cm segment of the duodenum that includes the duodenal bulb, i.e. Whipple procedure or similar
* Any histologically confirmed high grade dysplasia (HGD) or cancer, gastrointestinal bleeding and requirement for anticoagulation therapy after study start except for use of low dose aspirin
* Exclusion of patients utilizing strong a moderate inhibitors of CYP2D6 and CYP3A4
* Patients with evidence of human immunodeficiency virus (HIV) infection will be excluded from the study even if the HIV viral load is undetectable on suppressive therapy. Many of the HIV suppression anti-viral medications are moderate/strong inhibitors of CYP2D6 and CYP3A4 and are exclusions based on above
* Patients with evidence of chronic hepatitis B virus (HBV) or C virus (HCV) infection will be excluded from the study, even if the HBV/HCV viral load is undetectable on suppressive therapy. Many of the HBV/HCV suppression anti-viral medications are moderate/strong inhibitors of CYP2D6 and CYP3A4 and are exclusions based on above
* Patients with active H. pylori infection that is untreated or refractory to standard antibiotic therapy
* Patients with prior history of peptic ulcers complicated by bleeding, New York Heart Association (NYHA) Classification II-IV, active autoimmune diseases, on anticoagulants at risk of bleeding or abnormal corrected QT interval (QTc) prolongation will also be excluded. Patients enrolled in this trial are status post colectomy (with either IPAA or IRA) and thus would not be expected to be at risk of diverticulitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-06-07 (Estimated); Primary Completion 2026-12-17 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Percent change in duodenal polyp burden | Baseline to 6 months
  Will be determined based on the sum of diameters from all polyps. Will be assessed by comparing upper gastrointestinal (GI) endoscopies respectively. Will be described using a two-sided 95% confidence interval and examined for difference from zero with a one-side paired t-test.
Incidence of adverse events | Up to 7 months
  Will examine the proportion of patients with grade 2 or 3 adverse events according to the Common Terminology Criteria for Adverse Events version 5.0. Will be summarized as a proportion with a 1-sided 90% confidence interval.

SECONDARY OUTCOMES:
Percent change in rectal/pouch polyp burden | Baseline to 6 months
  Will be assessed by comparing the lower GI endoscopies. Results will be presented using summary statistics and corresponding confidence intervals.

OTHER OUTCOMES:
Percent change in immunohistochemical staining levels | Baseline to 6 months
  Will assess rectal and duodenal tissue samples for COX-2 expression level, beta-catenin, and Ki-67. Mean percent change in immunohistochemical staining levels will be associated with intestinal polyp burden using a scatterplot of the two variables and evaluated using a Spearman rank correlation statistic.
Proteomic profile | Baseline to 6 months
  Will identify proteins that are statistically significantly differently expressed between patients after treatment. The proteomic profile of serum will be correlated to clinical response to therapy and compared between baseline and end of intervention. No formal statistical inference will be performed. Proteins will be described with summary statistics to assist in planning follow-up studies.
TPST-1495 plasma concentrations | At pre-dose and 2-and 4-hours post-dose at 3 months visit
  Will assess steady-state pharmacokinetics.

CONTACTS AND LOCATIONS:
Overall Officials: Niloy J Samadder, Principal Investigator — University of Wisconsin Carbone Cancer Center - University Hospital
Locations (5):
- United States (4):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm